CLINICAL TRIAL: NCT02336880
Title: Short-term Internet-delivered Cognitive Behavioural Therapy for Treatment of Cardiac Anxiety and Fear of Body Sensations in Patients With Non-cardiac Chest Pain - a Pilot Randomized Controlled Study
Brief Title: Internet-delivered CBT for NCCP-patients - a Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Ostergotland County Council, Sweden (Other); Medical Research Council of Southeast Sweden (Other Government)
Responsible Party: Principal Investigator, Ghassan Mourad, Junior lecturer, PhD-student, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I-CBT in NCCP
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Chest Pain; Anxiety; Fear
MeSH Terms: conditions — Chest Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): 4 weeks guided internet-delivered cognitive behavioural therapy program. The program consists of psychoeducation, exposure to physical activity, and a breathing-based relaxation exercise
  Interventions: Behavioral: Internet-delivered cognitive behavioural therapy
- Control group (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: Internet-delivered cognitive behavioural therapy
  Arms: Intervention group

SUMMARY:
This pilot randomized controlled trial (RCT) aims to test the feasibility and effectiveness of a guided internet-delivered cognitive behavioural therapy intervention in the treatment of cardiac anxiety and fear of body sensations in patients with non-cardiac chest pain. The control group will receive care-as-usual.

DETAILED DESCRIPTION:
Despite reassurance, many patients with non-cardiac chest pain (NCCP) think they have an undetected cardiac disease and avoid activities that they think might be harmful to their heart. These patients need help and support to evaluate the way they perceive and handle their chest pain. Therefore, we have developed a 4 session guided intervention based on cognitive behavioural therapy that will be delivered via internet.

The intervention consists of psychoeducation, exposure to physical activity, and a breathing-based relaxation exercise. The goal with the intervention is to help the participants modify their beliefs about chest pain, change their cognitive and behavioural strategies, and give them tools to handle chest pain to prevent them from relapse.

ELIGIBILITY:
Inclusion Criteria:

* recurrent chest pain that has been diagnosed as non-cardiac at least twice during last 6 months
* patients screened positive for avoidance of physical activity due to cardiac anxiety and/or fear of body sensations

Exclusion Criteria:

* no regular access to a computer/tablet computer with internet connection
* language difficulties
* not able to perform physical activity/exercise test due to physical constraints
* patients with severe depressive symptoms
* patients with acute ischemic heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cardiac anxiety (Data collection) | 12 months
  Data collection will be performed before and after the intervention, and 3 and 12 months after the end of the intervention

SECONDARY OUTCOMES:
Fear of body sensations (Data collection) | 12 months
  Data collection will be performed before and after the intervention, and 3 and 12 months after the end of the intervention
Depressive symptoms (Data collection) | 12 months
  Data collection will be performed before and after the intervention, and 3 and 12 months after the end of the intervention
Healthcare utilization and costs (Data collection) | 12 months
  Data collection will be performed12 months after the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tiny Jaarsma, Professor, Study Chair — Linkoeping University
Locations (1):
- Linkoeping University, Linköping, Sweden

REFERENCES:
- [Derived] Mourad G, Stromberg A, Jonsbu E, Gustafsson M, Johansson P, Jaarsma T. Guided Internet-delivered cognitive behavioural therapy in patients with non-cardiac chest pain - a pilot randomized controlled study. Trials. 2016 Jul 26;17(1):352. doi: 10.1186/s13063-016-1491-1. PMID 27456689